CLINICAL TRIAL: NCT02496845
Title: An Open Label Randomized Study to Examine the Safety and Clinical Efficacy of Local Topical Dual Active Preparation for Erectile Dysfunction
Brief Title: Safety and Clinical Efficacy of Local Topical Treatment for Erectile Dysfunction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VasoLead (2012) Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VL#FIA3-30 #002
Record Dates: First submitted 2015-06-18; First posted 2015-07-14 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Topical treatment and PK. Administration of VL#FIA3-30 (dual administration of MH30-01 & IS045-01)
  Interventions: Drug: VL#FIA3-30
- Groups B, C, D (Experimental): Dual topical biweekly administration and intraurethral. Triple topical weekly administration. Multiple topical administration. Administration of VL#FIA3-30 (dual administration of MH30-01 & IS045-01)
  Interventions: Drug: VL#FIA3-30

INTERVENTIONS:
Drug: VL#FIA3-30 — Vasoactive dual treatment (MH30-01 & IS045-01)
  Other Names: Transdermal application

SUMMARY:
VL#FIA3-30 is a preparation intended for topical use, applied on the penis, for the treatment of ED.

DETAILED DESCRIPTION:
VasoLead's preparation to treat erectile dysfunction (ED), VL#FIA3-30, is composed of 2 active pharmaceutical ingredients, both act as vasodilators via different mechanisms. Both are currently used orally in the USA and Europe for the treatment of hypertension, angina pectoris and other diseases.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* ED for more than six months in duration.
* IIEF-EF domain score at baseline from 11 to 19 .
* Willingness for a minimum of two sexual attempts during the short period of this study.
* At least 50% unsuccessful sexual intercourse for 4 attempts on 4 different days.
* A stable heterosexual relationship with the same partner for more than six months.
* Age 25 to 75 years old.

Exclusion Criteria:

* Neurological pathology;
* Prior radical prostatectomy;
* Any unstable medical or psychiatric condition, spinal cord injury, or penile anatomical abnormalities;
* Clinically significant chronic hematological disease;
* Cardiovascular conditions that prevent sexual activity (CHF or severe coronary artery disease);
* History of myocardial infarction, stroke, or life-threatening arrhythmia within 6 months prior to enrollment into the study;
* Use of anti-androgens, or oral or injectable androgens;
* Documented hypotension (BP below 100 systolic or 70 diastolic) or known orthostatic hypotension;
* Routine use of more than 2 antihypertensive medications;
* Use of oral nitrates within 3 months prior to enrollment into the study;
* Cancer within the last 3 years;
* Documented allergic reaction;
* Investigators impression for patient non-compliance;
* Hepatic or renal failure;
* History of HIV, hepatitis B, hepatitis C;
* Is an immediate family member of personnel directly affiliated with the study at the investigative site, or is personally directly affiliated with the study at the investigative site;
* Subject has taken any investigational medication within 30 days prior of entry into the study
* Employed by VasoLead (2012) Ltd.

Ages: 25 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-11 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as a aeasure of safety and tolerability of topical VL#FIA3-30 applied on the penis | 2 weeks

SECONDARY OUTCOMES:
Increase the score level of the Erection Hardness Score (EHS) index | 2 weeks
Increase points of the International Index of Erectile Function-Erectile Function (IIEF-EF) score | 2 weeks
Significant increase of Flow Mediated Dilation (FMD) parameters | 2 weeks
Increase the total ED inventory of Treatment Satisfaction (EDITS) score | 2 weeks
Improvement of patient/Investigator satisfaction VAS score | 2 weeks
Increase the total score of the Quality of Erection Questionnaire (QEQ) | 2 weeks
Increase the total score of the modified Quality of Erection Questionnaire (mQEQ) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gruenwald Ilan, Prof., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel